CLINICAL TRIAL: NCT03681899
Title: Evaluation of Rupture of Galenic Practices at Home in a Population Aged 65 or Older
Acronym: CRUSHAGE
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH3-07
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2019-10

CONDITIONS: Geriatric Assessment
Keywords: Rupture of galenic; Ederly patients; Geriatry; Drug class
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects aged of 65 years or older: Subjects aged of 65 years or older, taking at least one oral medication for two weeks or more.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — * Socio-demographic data (age, sex, place of residence, and family status, last occupation, existence or not of a primary caregiver (family and / or professional));
  * Medical and surgical history (Charlson Comorbidity Scale);
  * Assessment of oral/dental condition
  * Record of drug treatments (number of oral medications per day, therapeutic class, number of daily intakes);
  * Oral treatments intake modalities (galenic breakdown of one or more drugs, usual or occasional, modalities of rupture, person responsible for the drugs, mixing with food / drink);
  * Autonomy evaluation (Lawton and Katz scales);
  * Mobility assessment (anamnestic evaluation);
  * Evaluation of Thyme (GDS 4 items);
  * Psycho-behavioral disorders,
  * Assessment of swallowing (presence of a diagnosis of dysphagia or suspicion based on anamnestic data).

SUMMARY:
Elderly people frequently take several medications and are exposed to iatrogenic risks.

The oral route is the preferred route of administration. The effectiveness and the safety of the drugs depend in particular on the modes of administration (frequency of the intake, respect of the doses and the galenic ...).

However, these modalities are very little known concerning the treatments intake at home in the elderly population.

In a health facility welcoming geriatric patients, the rupture of galenic is frequent and favored by swallowing disorders, dependence, the increase in age, the presence of cognitive disorders or psycho-behavioral disorders.

The consequences of the rupture of galenic are numerous, concern the patients but also the caregivers who administer the treatments.

DETAILED DESCRIPTION:
Primary objective :

- Estimate the rupture of galenic prevalence of at least one molecule in a population of subjects aged 65 years or over living at home and taking at least one oral drug for 2 weeks or more.

Secondary objectives:

* Identify the drug classes most frequently involved in the rupture of galenic in a population of subjects aged 65 years of age or over at home;
* Identify the actors of the drug administration in a population of subjects aged 65 years of or over at home;
* To determine the medical and sociodemographic factors associated with the rupture of galenic in a population of subjects aged 65 years or over at home;
* To determine the modalities of rupture of galenic in a population of subjects aged 65 or over at home.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 65 or over;
* Patient taking at least one oral medication for two weeks or more;
* Patient affiliated to a social security scheme;
* Patient who has agreed to reply to the questionnaire or, in case of inability to agree, agreement obtained from the caregiver or guardian/curator.

Exclusion Criteria:

* Patient unable to answer questionnaires and without a referent caregiver capable of reply ;
* Patient having changed residence for two weeks or less;
* Patient residing in a residential care facility for dependent elderly people.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient taking at least one oral medication for two weeks or more, regarless of the pathology.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Estimate the rupture of galenic prevalence of at least one molecule in a population of subjects aged 65 years or over living at home and taking at least one oral drug for 2 weeks or more. | 12 months
  Calculation of the prevalence of galenic rupture by dividing the number of persons with at least one rupture of galenic by the number of persons included in the study.

SECONDARY OUTCOMES:
To determine the drug classes most frequently involved in the rupture of galenic in a population of subjects aged 65 years of age or over at home | 12 months
  Number of participants for each drug class
To determine the drug classes most frequently involved in the rupture of galenic in a population of subjects aged 65 years of age or over at home | 12 months
  Percentage of participants for each drug class
To determine the actors of the drug administration in a population of subjects aged 65 years of or over at home | 12 months
  Number of participants for each actor
To determine the actors of the drug administration in a population of subjects aged 65 years of or over at home | 12 months
  Percentage of participants for each actor
To determine the medical and sociodemographic factors associated with the rupture of galenic in a population of subjects aged 65 years or over at home | 12 months
  Binary logistic regression with variable to explain, the rupture of galenic
To determine the medical and sociodemographic factors associated with the rupture of galenic in a population of subjects aged 65 years or over at home | 12 months
  Binary logistic regression with variable as explanatory variables, the medical and sociodemographic factors
To determine the modalities of rupture of galenic in a population of subjects aged 65 or over at home | 12 months
  Number of paticipants for each modality
To determine the modalities of rupture of galenic in a population of subjects aged 65 or over at home | 12 months
  Percentage of paticipants for each modality

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique, France

IPD SHARING:
Plan to Share IPD: No